CLINICAL TRIAL: NCT01770548
Title: Autism and Glutamatergic Synapse : Research of Genetic Mutations and Identification of Clinical and Neurophysiological Markers.
Brief Title: Neurophysiological Molecular and Developmental Analysis of the Glutamate Synapse in Autism
Acronym: NMDA-Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: AORT08-FBB/NMDA-Autism; 2008-A01162-53 (Other: ID RCB)
Record Dates: First submitted 2013-01-15; First posted 2013-01-17 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder | interventions — Evoked Potentials, Auditory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Autism (Experimental): Analysis of the glutamate synapse in autism
  Interventions: Genetic: analysis of the glutamate synapse in autism; Genetic: DNA collection; Other: Auditory evoked potentials
- Relative (Other): Analysis of the glutamate synapse in autism
  Interventions: Genetic: analysis of the glutamate synapse in autism; Genetic: DNA collection; Other: Auditory evoked potentials
- Major control (Other): DNA collection
  Interventions: Genetic: analysis of the glutamate synapse in autism; Genetic: DNA collection; Other: Auditory evoked potentials
- Minor control (Other): auditory evoked potentials
  Interventions: Other: Auditory evoked potentials

INTERVENTIONS:
Genetic: analysis of the glutamate synapse in autism — Neurophysiological, molecular and developmental analysis of the glutamate synapse in autism
  Arms: Autism; Major control; Relative
Genetic: DNA collection — DNA collection
  Arms: Autism; Major control; Relative
Other: Auditory evoked potentials — auditory evoked potentials

SUMMARY:
Neurophysiological, Molecular and Developmental Analysis of the glutamate synapse in Autism

DETAILED DESCRIPTION:
Analysis about 50 genes in glutamate synapse

ELIGIBILITY:
Inclusion Criteria:

* have a Pervasive Developmental Disorder

Exclusion Criteria:

* N/A

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 497 (Actual)
Dates: Start 2009-01; Primary Completion 2011-01 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
screening of about 50 genes encoding proteins of the NMDA receptor complex, chosen according to their chromosomal localisation located in hotspots depicted by genome-wide screens in large population of autistic patients | two years

CONTACTS AND LOCATIONS:
Overall Officials: Frédérique BONNET-BRILHAULT, MD PHD, Study Director — University François Rabelais of TOURS
Locations (4):
- France (4):
  - CHRU - Centre de Ressources Autisme (CRA), Brest
  - CHS du ROUVRAY, Rouen
  - Chru - Cic, Tours
  - CHRU - Pédopsychiatrie, Tours

REFERENCES:
- [Result] Bonnet-Brilhault F, Alirol S, Blanc R, Bazaud S, Marouillat S, Thepault RA, Andres CR, Lemonnier E, Barthelemy C, Raynaud M, Toutain A, Gomot M, Laumonnier F. GABA/Glutamate synaptic pathways targeted by integrative genomic and electrophysiological explorations distinguish autism from intellectual disability. Mol Psychiatry. 2016 Mar;21(3):411-8. doi: 10.1038/mp.2015.75. Epub 2015 Jun 9. PMID 26055424